CLINICAL TRIAL: NCT04012229
Title: IMpact of BrcA Status on Survival in Adjuvant Breast Cancer (IMBASSA)
Brief Title: IMpact of Breast cAncer Gene Status on Survival in Adjuvant Breast Cancer (IMBASSA)
Acronym: IMBASSA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/291
Record Dates: First submitted 2019-04-29; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; BRCA1 Mutation; BRCA2 Mutation
Keywords: Breast cancer; BRCA1; BRCA2; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated by chemotherapy for an early breast cancer: Patients (Women or Men) older than 18 years old, histologically confirmed invasive early breast cancer, treated by neo-adjuvant and/or adjuvant chemotherapy with the first cure of chemotherapy received between January 1st, 2003 and December 31th, 2013 were included.
  Interventions: Genetic: BRCA mutation

INTERVENTIONS:
Genetic: BRCA mutation — The genetic testing was performed according interregional consensus (Manchester score > or = 16) on blood sample using classical chain-termination (Sanger sequencing) and multiplex ligation-dependant probe amplification to search large rearrangements.

SUMMARY:
Relationship between the presence of the BRCA mutation (BReast Cancer) and outcomes is unclear in high-risk early breast cancers (BC).

This study is a multi-center retrospective cohort of patients treated in region Franche-Comté for an early BC by neoadjuvant and/or adjuvant chemotherapy.

The primary aim was to describe clinical and pathological characteristics considering BRCA mutated (BRCAm) patients versus BRCA wild type (BRCAwt) patients or untested patients. The second objective was to assess the prognostic impact of germinal BRCAm in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old,
* Histologically confirmed invasive early breast cancer
* Neo-adjuvant and/or adjuvant chemotherapy with the first cure of chemotherapy received between January 1st, 2003 and December 31th, 2013

Exclusion Criteria:

* Clinical, radiological or histological confirmed metastatic disease
* Non-invasive breast cancer,
* Patients who received incomplete treatment
* Patients who did not speak French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated in region Franche-Comté, France, for an early breast cancer, by neoadjuvant and/or adjuvant chemoterapy.
  Eight center were included : University hospital of Besançon, Polyclinique de Franche-Comté (Besançon), Clinique Saint-Vincent (Besançon), Hospitals of Vesoul, Lons-le-Saunier, Pontarlier, Dole and Montbéliard.
Sampling Method: Non-Probability Sample
Enrollment: 2295 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Age of diagnosis | one day
  The date from the date of birth to the date of pathological diagnosis (Years)
Pathological tumor size | one day
  Pathological tumoral size after partial or complete surgery
  Pathological size in millimeters after complete surgery
Pathological nodal involvement | one day
  Presence of metastasis on complete lymphadenectomy
Clinical tumor size | one day
  Clinical measurement of the tumor in millimeters after surgery
Clinical nodal involvement | one day
  Presence of axillary lymph nodes before surgery (no versus yes)
Estrogen receptor expression status | one day
  Expression of estrogen receptors on tumor after surgery (% expression in immuno-histo-chemistry, ranging from 0 to 100%.
Progesterone receptor expression status | one day
  Expression of progesterone receptor on tumor after surgery (% expression in immuno-histo-chemistry, ranging from 0 to 100%.
HER2 status | one day
  Expression of HER2 on tumor after surgery (expression assessed by immuno-histo-chemistry, if HER2 is ++, fluorescence in situ hybridization. HER2 status is ranged to not overexpressed (0 and +), equivocal (++) and overexpressed (+++).
Sexe | one day
  Male or Female
Scarff Bloom and Richardson grade (SBR) | one day
  This grade is the addition of score of tubule formation (>75% 1 point 10%-75% 2 point <10% 3 points), nuclear pleomorphism (small, regular uniform cells 1 point moderate increase in size and variability 2 points, marked Variation 3 points) and mitotic counts (dependent on microscope field area 1-3 points) assessed by pathology analysis on tumor after surgery. The SBR grade is ranging from I (total of 3 to 5), II (6 and 7) and III (8 and 9).
In situ component | one day
  Presence or absence of in situ carcinoma assessed by pathology analysis on tumor after surgery
Pathological histotype | one day
  Histologic subtype of breast tumor : ductal, lobular or other, assessed by pathology analysis on tumor after complete surgery
Metastatic sites (if available) | one day
  Metastatic sites of primary breast cancer : Nodal (other than axillary), lung, liver, bone, cerebral and other sites.
Medical treatment | one day
  Type of chemotherapy (adjuvant, neoadjuvant, metastatic)

SECONDARY OUTCOMES:
Overall Survival | one day
  The time from the date of first treatment or of first consultation, whichever comes first, to the date of death from any cause.
Invasive Disease Free Survival | one day
  The time from the date of the first treatment or th first consultation to the date of local or ipsilateral or controlateral invasive breast cancer, or other invasive cancer or distant recurrence or death from breast cancer or any cause
Distant Disease Free Survival | one day
  The time from the date of the first treatment or the first consultation to the date of distant recurrence or death from breast cancer or any cause

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Jean Minjoz, Besançon, Franche-Comté, France